CLINICAL TRIAL: NCT01420705
Title: The Effect of Giving BCG Vaccine at Birth to Low Birth-weight Infants on Development of Allergy and Asthma in Childhood - Follow up of a Randomised Trial in Guinea-Bissau
Brief Title: Bacille Calmette-Guérin (BCG) Vaccine and Atopy
Status: Completed | Type: Observational
Sponsor: Bandim Health Project (Other)
Collaborators: Murdoch Childrens Research Institute (Other)
Responsible Party: Peter Aaby, Bandim Health Project
Other Study IDs: 2011-BHP-LBW-BCG-atopy
Record Dates: First submitted 2011-08-12; First posted 2011-08-22 (Estimated); Last update posted 2011-12-29 (Estimated); Status verified 2011-12

CONDITIONS: Asthma; Eczema; Food Hypersensitivity
Keywords: Bacille Calmette-Guérin; DTP; Vaccination; Allergy; Atopy; Guinea-Bissau
MeSH Terms: conditions — Asthma; Eczema; Food Hypersensitivity; Hypersensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Faecal samples are collected for analyses of parasites and microbes
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Low birth-weight cohort: Children previously enrolled in randomised trial NCT00146302 who are currently living within the Bandim Health Project study area

SUMMARY:
The prevalence of asthma and allergic diseases is increasing worldwide. Infections and vaccinations in childhood may have an impact on the subsequent development of asthma and allergy. In Guinea-Bissau, the investigators previously found that Bacille Calmette-Guérin (BCG) vaccine was associated with reduction in atopy. Since then the investigators have conducted a randomised trial of BCG vaccine given at birth to low birth-weight infants. The present study aims to follow up children enrolled in the BCG randomised trial to assess for asthma and allergy later in childhood. Based on previous observations, the investigators expect children allocated to receive BCG at birth will have a reduction in allergy profile when compared to children who did not receive BCG at birth.

DETAILED DESCRIPTION:
Background: Prevalence of asthma and allergy is increasing worldwide, and the cause is unclear. Previous work by the Bandim Health Project and others has identified that infections and routine childhood vaccinations have an impact on the development of atopic sensitisation and allergic symptoms later in life. A number of these studies have found association between BCG vaccination and reduction in atopy and allergy. Only one randomised trial has been conducted of BCG vaccine to protect against allergy with inconclusive results. The present project provides the opportunity to follow-up children born low birth-weight who were randomised to receive BCG vaccine at birth or to receive BCG later in infancy as part of regular care.

Hypothesis:

* Children given BCG vaccine at birth will have reduced prevalence of positive skin-prick test and allergic symptoms when compared with children who did not receive BCG at birth
* Early BCG vaccination will be associated with reduced prevalence of positive skin prick test and allergic symptoms
* Early DTP vaccination will be associated with increased prevalence of positive skin-prick tests and allergic symptoms

Objectives:

* to examine the effects of environmental factors, including BCG, DTP and measles vaccines, on atopy (determined by skin-prick tests) and symptoms of asthma, eczema and food allergy
* to examine the sex-differential effects of vaccination on atopy and allergic symptoms
* to determine the association between faecal microbial diversity, atopy and food allergy

Methods: children previously enrolled in NCT00146302 will followed up at home (currently aged 3-9 years) and tested for atopic sensitisation with skin-prick tests and presence of allergic symptoms determined by questionnaire.

Sample size: 812 children from the Bandim Health Project study area were enrolled in the randomised trial. The investigators anticipate to be able to follow up approximately 487 of these children, which will have the power to detect a 30% difference in atopic sensitisation between groups.

ELIGIBILITY:
Inclusion Criteria:

* Previous enrolment in NCT00146302
* Living within Bandim Health Project study area

Exclusion Criteria:

* Children with known history of anaphylaxis
* Children with skin infections or severe skin conditions for who SPT could not be reliably performed
* Children currently taking anti-histamine medication

Ages: 3 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children previously enrolled in NCT00146302 living within Bandim Health Project study area, Bissau
Sampling Method: Probability Sample
Enrollment: 487 (Estimated)
Dates: Start 2011-10; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Skin prick test | Single observation at time of consent - DAY 1
  Skin prick tests to common aero and food allergen

SECONDARY OUTCOMES:
Symptoms of asthma | Single observation at time of consent - DAY 1
  Symptoms of asthma using questions modified from ISAAC
Symptoms of eczema | Single observation at time of consent - DAY 1
  Eczema symptoms using questions modified from ISAAC
Symptoms of food allergy | Single observation at time of consent - DAY 1
  Symptoms of food allergy using questions modified from the Health Nuts study

CONTACTS AND LOCATIONS:
Overall Officials: Peter Aaby, DMSc, Principal Investigator — Bandim Health Project
Locations (1):
- Bandim Health Project, Bandim, Guinea-Bissau

REFERENCES:
- [Derived] Kiraly N, Benn CS, Biering-Sorensen S, Rodrigues A, Jensen KJ, Ravn H, Allen KJ, Aaby P. Vitamin A supplementation and BCG vaccination at birth may affect atopy in childhood: long-term follow-up of a randomized controlled trial. Allergy. 2013 Sep;68(9):1168-76. doi: 10.1111/all.12216. Epub 2013 Aug 31. PMID 23991838
- See also: Related Info — http://www.bandim.org